CLINICAL TRIAL: NCT05979779
Title: A 6-Month, Randomized, Double-Blind, Placebo-controlled, Phase 2 Study of the Safety and Efficacy of Three HU6 Dose Levels and Placebo in Nonalcoholic Steatohepatitis
Brief Title: Ph 2 Study of the Safety and Efficacy of Three HU6 Dose Levels and Placebo in Nonalcoholic Steatohepatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-HU6-2202
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, randomized, parallel-group, placebo-controlled, double-blind study where subjects will be randomized to one of 3 HU6 dose levels or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment: HU6 Planned doses of HU6 (Experimental)
  Interventions: Drug: HU6
- Placebo Comparator Non-active study drug (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HU6 — HU6 is being evaluated for its efficacy in improving liver fat content in subjects with Nonalcoholic Steatohepatitis (NASH)
  Arms: Active Treatment: HU6 Planned doses of HU6
Other: Placebo — Placebo
  Arms: Placebo Comparator Non-active study drug

SUMMARY:
This is a phase 2 randomized, double-blind, placebo-controlled parallel group study of 3 dose levels of HU6 in subjects with nonalcoholic steatohepatitis (NASH). Six months (26 weeks) of dosing is planned, and subjects will be followed for safety, efficacy, pharmacodynamics (PD), and pharmacokinetics (PK) during this time. The end-of-study visit will take place approximately 4 weeks after the last dose of the study drug (Week 30).

DETAILED DESCRIPTION:
This is a phase 2 randomized, double-blind, placebo-controlled parallel group study of 3 dose levels of HU6 (150 mg, 300 mg, and 450 mg) and placebo in approximately 204 subjects with NASH.

Subjects will be screened over a 49-day period to determine their eligibility based on specific history, physical, laboratory, and imaging evaluations, which will require more than one visit during the screening period. On Day 1, subjects will be randomized 2:1:2:2 into 1 of 4 treatment groups (placebo, 150 mg HU6, 300 mg HU6, or 450 mg HU6). Six months (26 weeks) of dosing is planned, and subjects will be followed for safety, efficacy, PD, and PK during this time. The end-of-study visit will take place approximately 4 weeks after the last dose of the study drug (Week 30).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the procedures and requirements of the study and provide written informed consent and authorization for protected health information disclosure.
2. Willing and able to comply with the requirements of the study protocol.
3. Male or female ≥18 years of age at time of informed consent.
4. Subject has a screening Fibroscan® CAP score >306 decibels per meter (dB/m) and interquartile range to median ratio (IQR/Med) <30%.
5. Subject has ≥8% liver fat determined by screening Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF).
6. Subject has moderate to advanced liver fibrosis based on documented history of biopsy score of F2 or F3 within 12 months prior to Screening, or subject has a screening Fibroscan® vibration-controlled transient elastography (VCTE) score ≥ 7.0 to ≤ 15.0 kPa.
7. Body mass index (BMI) ≥27.0 kg/m2.
8. Clinically euthyroid as assessed by a thyroid profile utilizing TSH and T4 testing at screening as assessed by the investigator based on the medical history of the subject.
9. Subjects with a diagnosis of glaucoma must be controlled and stable (no changes in treatment regimen within 3 months prior to Screening).
10. Inclusion as per investigator assessment of general medical status and as documented by medical history, physical examination, vital sign assessments, 12-lead ECG, clinical laboratory assessments, and general observations.

Exclusion Criteria:

Subjects will be excluded from the study if any of the following criteria are met:

1. The subject has a history of cirrhosis and/or hepatic decompensation, including ascites, hepatic encephalopathy, or variceal bleeding.
2. The subject has a history of acute pancreatitis within 1 year of Screening or chronic pancreatitis of any cause.
3. History of any bariatric surgery intervention, including but not limited to lap banding, intragastric balloon, duodenal-jejunal sleeve, or bariatric surgery or plans for bariatric surgery prior to conclusion of study participation.
4. Have obesity induced by other endocrinologic disorders (e.g., Cushing Syndrome, polycystic ovarian syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome).
5. Any surgical or medical condition or history that, in the opinion of the investigator in consultation with the medical monitor, may potentially alter the absorption, metabolism, or excretion of study treatment.
6. History of or treatment for clinically significant gastroparesis, inflammatory bowel disease, or any surgery of the upper gastrointestinal tract with the exception of cholecystectomy, or minor gastric procedures that are approved by the medical monitor.
7. History (including any family history) of malignant hyperthermia.
8. History of chronic serious recurrent skin rashes of unknown cause.
9. History of malignancy within 5 years (except cutaneous basal or squamous cell carcinoma, carcinoma-in-situ, or low-grade prostate cancer).
10. History of the following cardiovascular conditions within 3 months prior to randomization: acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, hospitalization due to congestive heart failure (CHF), or acute CHF.
11. NYHA Functional Class II, III, or IV heart failure.
12. Subject has a pacemaker.
13. Active kidney disease requiring therapy, kidney transplant, or eGFR <45 mL/min/1.73 m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation.
14. Significant and unstable lung disease (chronic obstructive pulmonary disease [COPD], emphysema, pulmonary fibrosis, or asthma) requiring oxygen or chronic daily medication. Note that mild, stable COPD and asthma on inhalers are allowed.
15. Subject has a diagnosed history of obstructive sleep apnea or uses continuous positive airway pressure (CPAP).
16. Subject has a history of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to Screening.
17. Subject has any history of agranulocytosis.
18. Subject has Wilson's disease.
19. Familial (mother/father/sibling) and/or personal history of retinal detachment any time in the past.
20. Subject has history of prior vitrectomy due to prior retinal condition.
21. Subject has a contraindication to dilation for ophthalmologic examination.
22. Evidence of the following on screening ophthalmologic examination:

    1. Peripheral retinal pathology, retinal tears, lattice, or nondiabetic ocular condition that requires treatment or intervention within 3 months of Screening.
    2. Diabetic retinopathy with macular exudates or macular edema (evidence of microaneurysms is not an exclusion).
    3. Any active macular disease that affects the vision, including macular pucker (epiretinal membrane), retinal vein occlusion, and macular degeneration.
    4. Subjects with significant visual impairment due to lens opacity from cataracts such that surgery will be required within the duration of the study in the opinion of the consulting ophthalmologist. (Subjects with cataract surgery >3 months prior to Screening may be included.)
    5. Subject has substantial media opacities that preclude successful retinal imaging.
23. Any condition (e.g., ongoing substance, drug, or alcohol abuse) that may interfere with participation or safety of investigations, in the opinion of the Investigator.
24. A history of moderate alcohol consumption defined as drinking ≥ 2 drinks per day for men or ≥ 1 drink per day for women. (A drink is defined as 12 ounces of beer, 5 ounces of wine, 1.5 ounces of distilled spirits.).
25. Subjects with untreated, uncontrolled, or unstable hypertension (systolic blood pressure [SBP] >160 and/or diastolic blood pressure [DBP] >100 mmHg upon repeat evaluation at screening). If subject is treated with antihypertensive medication, the regimen must be stable at least 1 month prior to screening.
26. Subjects with untreated or persistent hypotension (SBP <90 mmHg) or symptomatic hypotension (that, in the opinion of the Investigator, requires active treatment).
27. Tachycardia (>100 beats/minute) at screening.
28. QTcF > 450 msec at screening for males and QTcF > 470 msec at screening for females.
29. Use of any of the following medications:

    1. The following oral antidiabetic drugs are prohibited within 3 months prior to screening and continuing throughout the study: insulin, meglitinides, thiazolidinediones, glucagon-like peptide (GLP-1) agonists, and gastric inhibitory polypeptide (GIP)/GLP-1 agonists.
    2. The following are prohibited within 3 months prior to screening (or planned use during the study) when used for weight loss: herbal preparation, over the counter (OTC) drug, mail order or prescription drug.
    3. Prescription or OTC stimulants including: dextroamphetamine/Dexedrine, dextroamphetamine/amphetamine combination product/Adderall, or methylphenidate (Ritalin®, Concerta®).
    4. Recent (within 3 months of screening) or current use of obeticholic acid/Ocaliva, systemic corticosteroids, methotrexate, tamoxifen, amiodarone, or long-term use of tetracyclines.
    5. Warfarin, heparin, factor Xa inhibitors (e.g., dabigatran, betrixaban, edoxaban, apixaban, and rivaroxaban).
    6. Vitamin E: use of ursodiol or high-dose vitamin E (>400 IU/day) for at least 1 month within the previous 6 months or started high dose vitamin E within the previous 3 months of Screening.
    7. Drugs with high risk of idiosyncratic drug-induced neutropenia (IDIN) or agranulocytosis (Andres 2018, Curtis 2017): antithyroid drugs (propylthiouracil and methimazole), ticlopidine, clozapine, phenothiazines, sulfasalazine, vancomycin, amoxicillin, ceftriaxone, ciprofloxacin, cotrimaxozole, piperacillin-tazobactam, and trimethoprim-sulfamethoxazole (Bactrim® or Septra®).
    8. Concomitant medications that prolong the QT/QTc interval and are known to be associated with increased risk of Torsade des pointes as identified in the https://crediblemeds.org/ website list category of 'Known Risk.'
30. Have acute or chronic hepatitis, signs, and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD)/NASH, or any of the following, as determined by the central laboratory during screening:

    1. International normalized ratio (INR) ≥1.3, or
    2. ALT >5.0× the ULN for the reference range, or
    3. AST >5.0× the ULN for the reference range, or
    4. Alkaline phosphatase (ALP) >2.0× the ULN for the reference range, or
    5. Total bilirubin >1.2× the ULN for the reference range (except for cases of known Gilbert's Syndrome).
31. Laboratory Values at Screening:

    1. Hemoglobin <9.5 g/dL, or
    2. ANC ≤1500/μL, or
    3. Marked hypertriglyceridemia (>1000 mg/dL), or
    4. Copper <LLN for the reference range, or
    5. Ceruloplasmin <LLN for the reference range, or
    6. Serologic evidence of hepatitis B based on hepatitis B surface antigen (HBsAG), or
    7. Serologic evidence of hepatitis C antibody (HCV Ab) and HCV RNA, or
    8. Serologic evidence of human immunodeficiency virus (HIV).
    9. Hemoglobin A1c (HbA1c) > 9.5%.
32. Intolerance to MRI or with conditions contraindicated for MRI procedures including but not limited to:

    1. Having surgical clips/metallic implants/shrapnel -or-
    2. Claustrophobia, have a history of claustrophobia, or intolerance of closed or small spaces.
33. Participation in another clinical trial at the time of screening or exposure to any investigational agent, including topical agents, within 30 days or 5 half-lives prior to Day 1, whichever is longer.
34. For subjects with a recent active viral, bacterial, or parasitic infection, they must have discontinued any treatment for their infection at least 5 days prior to screening. Patients who test positive for COVID-19 during the screening period must have a negative rapid antigen test prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in liver fat, as assessed by magnetic resonance imaging liver proton density fat fraction (MRI-Liver PDFF) at 6 months (26 weeks) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rob Schott, MD, Study Director — Rivus Pharmaceuticals, Inc.
Locations (20):
- United States (20):
  - ProSciento CRU, Chula Vista, California
  - Velocity Clinical Research, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Northern California Research Center, Sacramento, California
  - Metro Clinical Trials, San Bernardino, California
  - Synergy Healthcare, Bradenton, Florida
  - ABMED Clinical Research Corp., Cape Coral, Florida
  - Southwest General Healthcare Center, Fort Myers, Florida
  - Miami Clinical Research, Miami, Florida
  - Advanced Clinical Research, Miami, Florida
  - Century Research, LLC, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - CenExel HRI, Berlin, New Jersey
  - Lillestol Research, Fargo, North Dakota
  - IMA Clinical Research-Austin, Austin, Texas
  - Mt Olympus Medical Research, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No